CLINICAL TRIAL: NCT02640716
Title: The Cog-VACCINE Study: a Randomized Controlled Clinical Trial to Evaluate the Effect of Cognitive Training in Patients With Vascular Cognitive Impairment, no Dementia
Brief Title: Cog-VACCINE: Cognitive Training in Patients With Vascular Cognitive Impairment, no Dementia
Acronym: Cog-VACCINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yi Tang, Dr., Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015010
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Vascular Cognitive Impairment no Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- training group (Active Comparator): Intervention: Multi-domain adaptive internet-based training program, including processing speed, attention, long-term memory, working memory, flexibility, calculation, and problem solving. 5 x 30 minutes per week, for 7 weeks.
  Interventions: Behavioral: multi-domain internet-based adaptive training program
- control group (Placebo Comparator): Intervention: placebo program: a fixed, primary difficulty level task. 5 x 30 minutes per week, for 7 weeks.
  Interventions: Behavioral: placebo program

INTERVENTIONS:
Behavioral: multi-domain internet-based adaptive training program — The cognitive training will be a multi-domain adaptive training program, including processing speed, attention, long-term memory, working memory, flexibility, calculation, and problem solving. Specific training paradigms include a time perception task, visual search task, attention blink, delayed mapping task, attention span task, Go-No go task, Stroop task, task switching, and name-face match task, among others. To maintain task difficulty, the tasks will be grouped based on the task difficulty in each domain. Furthermore, each task will have various difficulty levels.
  Arms: training group
Behavioral: placebo program — For the control group, tasks for processing speed and attention are included. Importantly, a fixed, primary difficulty level for all participants in the control group is set.
  Arms: control group

SUMMARY:
This study evaluates the efficacy and mechanism of internet-based cognitive training in patients with subcortical VCIND. Half of participants will receive multi-domain adaptive internet-based training program, while the other half will receive a fixed, primary difficulty level task.

DETAILED DESCRIPTION:
Background:

Vascular cognitive impairment no dementia (VCIND) refers to cognitive deficits associated with underlying vascular causes which fall short of a dementia diagnosis. Because of its high prevalence and high progression to dementia, interest in VCIND has greatly expanded in recent years. Although it has been widely recognized that early intervention of VCIND holds the potential to delay or even reverse the cognitive impairment, no treatment is available yet. Executive dysfunction is the characteristic impairment in subcortical VCIND, and cognitive training significantly improved executive and other aspects of cognitive function in health older adults and patients with cognitive impairment. Whether and how cognitive training improves cognitive function in patients with VCIND remains largely unknown.

Objectives:

The primary objective of this double-blinded, randomized RCT is to assess whether internet-based cognitive training in patients with subcortical VCIND improves their cognitive abilities. The second objective is to evaluate the effect of cognitive training on neural plasticity, including brain activation and white matter integrity, which are assessed by functional and structural MRI. Finally, possible genetic and plasma biomarkers related to a positive effect or lack of effect of the training will be examined.

Patients and Methods:

The proposed study is a three-center, double-blinded, randomized controlled trial that will include 60 patients diagnosed with VCIND from the neurology clinics at Beijing Friendship hospital, Xuan Wu hospital, and geriatric clinic at Fu Xing hospital, Capital Medical University. The patients will be randomized to either a training or a control group. The intervention is internet-based cognitive training performed for 30 minutes over 35 sessions. Neuropsychological assessment and functional magnetic resonance imaging (MRI) will be performed before and 7 weeks after training.

Relevance:

Currently there is no known treatment available for VCIND. The proposed study is to determine the efficacy of cognitive training in patients with VCIND. Secondly, using functional and structural MRI, this study is to reveal the potential mechanism underlying cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Literate Han Chinese, aged 50-78 years, with a consistent caregiver who accompanies the subject at least 4 days a week;
* Complaint and/or informant report of cognitive impairment involving memory and/or other cognitive domains lasting for at least 3 months;
* Neither normal nor demented according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, with a clinical dementia rating (CDR) ≥ 0.5 on at least one domain and global score ≤ 0.5; a Mini-Mental State Examination (MMSE) score ≥ 20 (primary school) or ≥ 24 (junior school or above);
* Normal or slightly impaired activities of daily living as defined by a total score of ≤ 1.5 on the three functional CDR domains (home and hobbies, community affairs, and personal care).

The MRI entry criteria are as follows:

* Multiple (≥ 3) supratentorial subcortical small infarcts (3-20 mm in diameter), with/without white matter lesions (WML) of any degree; or moderate to severe WML (score ≥ 2 according to the Fazekas rating scale) with/without small infarct;
* Absence of cortical and watershed infarcts, hemorrhages, hydrocephalus, and WMLs with specific causes (e.g., multiple sclerosis);
* No hippocampal or entorhinal cortex atrophy (score 0 according to the medial temporal lobe atrophy scale of Scheltens).

Exclusion Criteria:

* severe aphasia, physical disabilities, or any other factor that may preclude completion of neuropsychological testing;
* disorders other than subcortical VCIND that may affect cognition;
* a Hamilton depression scale (HAMD) score >17 or schizophrenia;
* new strokes within 3 months before baseline;
* inherited or inflammatory small vessel disease;
* clinically significant gastrointestinal, renal, hepatic, respiratory, infectious, endocrine, or cardiovascular system disease;
* cancer, alcoholism, drug addiction;
* use of medications that may affect cognitive functioning, including tranquilizers, anti-anxiolytics, hypnotics, nootropics, and cholinomimetic agents;
* inability to undergo a brain MRI.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2017-05-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, M.D., Ph.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li QG, Xing Y, Zhu ZD, Fei XL, Tang Y, Lu J. Effects of computerized cognitive training on functional brain networks in patients with vascular cognitive impairment and no dementia. CNS Neurosci Ther. 2024 Jun;30(6):e14779. doi: 10.1111/cns.14779. PMID 38828650
- [Derived] Tang Y, Zhu Z, Liu Q, Li F, Yang J, Li F, Xing Y, Jia J. The efficacy of Cognitive training in patients with VAsCular Cognitive Impairment, No dEmentia (the Cog-VACCINE study): study protocol for a randomized controlled trial. Trials. 2016 Aug 5;17(1):392. doi: 10.1186/s13063-016-1523-x. PMID 27496126

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Training Group | Control Group
Started (Completed baseline assessments and randomized) | 30 | 30
Training Completion (Training completion) | 27 | 27
Completed (6-month follow-up) | 23 | 21
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.9) | 64.9 (6.6) | 64.4 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 18 | 22 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for cognitive dysfunction. It is rated on a 30-point scale and assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The higher score represents a better cognitive function.
  units on a scale | 21.9 (3.8) | 21.2 (3.8) | 21.5 (3.8)
Trail Making Test B-A (TMT B-A) [Mean (Standard Deviation); unit: second] — The Trail Making Test is a commonly used neuropsychological test of visual attention and task-switching. In two timed tasks, subjects are asked to first connect numbers (Test A), then alternating numbers and letters (Test B), in sequential order as quickly as possible. Completion times, relating to cognitive processing speed and executive function (respectively) are represented as a difference (B-A).
  second | 74.0 (56.6) | 77.0 (65.3) | 75.5 (60.5)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Mean Change of the Montreal Cognitive Assessment (MoCA)
Description: The study uses MoCA to assess changes in the global cognitive function after an intervention of cognitive training. Baseline and 7-week were the two relevant time points used in the calculation.
  The score of MoCA ranges from 0 to 30, and higher scores mean a better outcome.
Time Frame: Baseline and 7 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale | 3.356 [1.467 to 5.244] | -0.085 [-2.062 to 1.892]

2. Primary Outcome: Estimated Mean Change of the Trail Making Test (TMT) B-A
Description: The Trail Making Test is a commonly used neuropsychological test of visual attention and task-switching. In two timed tasks, subjects are asked to first connect numbers (Test A), then alternating numbers and letters (Test B), in sequential order as quickly as possible. Completion times, relating to cognitive processing speed and executive function (respectively) are represented as a difference (B-A). The Trail Making Test is a commonly used neuropsychological test of visual attention and task-switching. In two timed tasks, subjects are asked to first connect numbers (Test A), then alternating numbers and letters (Test B), in sequential order as quickly as possible. Completion times, relating to cognitive processing speed and executive function (respectively) are represented as a difference (B-A). The change from baseline at week 7 in the B-A difference is reported as a primar
Time Frame: Baseline and 7 weeks
Measure: Mean (95% Confidence Interval); unit: second
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 30 | 30
second | -5.958 [-38.558 to 26.642] | -10.702 [-45.259 to 23.856]

3. Secondary Outcome: Estimated Mean Changes in Left Hippocampal Volume
Description: The left hippocampal volume on structural Magnetic Resonance Imaging (MRI) was measured by voxel-based morphometrics. The estimated mean changes in left hippocampal volume from baseline at week 7 is reported.
Time Frame: Baseline and 7 weeks
Measure: Mean (95% Confidence Interval); unit: Cubic millimeter
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 30 | 30
Cubic millimeter | -105.673 [-287.585 to 76.239] | -70.266 [-269.430 to 128.899]

4. Secondary Outcome: Estimated Mean Change in Right Hippocampal Volume
Description: The right hippocampal volume on structural Magnetic Resonance Imaging (MRI) was measured by voxel-based morphometrics. The estimated mean change in right hippocampal volume from baseline at week 7 is reported.
Time Frame: Baseline and 7 weeks
Measure: Mean (95% Confidence Interval); unit: Cubic millimeter
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 30 | 30
Cubic millimeter | -0.276 [-185.672 to 185.119] | -103.716 [-316.408 to 108.975]

5. Secondary Outcome: Estimated Mean Change in Brain White Matter Integrity
Description: The white matter microstructure was measured by diffusion tensor imaging (DTI) . The whole-brain average fractional anisotropy (FA) was calculated to show brain white matter integrity. The change of whole-brain average FA from baseline at week 7 is reported.
  Fractional anisotropy (FA) is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions.
Time Frame: Baseline and 7 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 30 | 30
units on a scale | -0.008 [-0.031 to 0.014] | 0.004 [-0.015 to 0.023]

6. Other Pre Specified Outcome: Estimated Mean Change of MoCA
Description: The participants will be followed up 6 months after recruitment. The training is not mandatory after 7 weeks, but the training details will be acquired from the online system. The change from baseline at month 6 in the MoCA difference is reported.
  The score of Moca ranges from 0 to 30, and higher scores mean a better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale | 2.224 [0.256 to 4.192] | 1.358 [-0.899 to 3.614]

ADVERSE EVENTS:
Time Frame: 7 weeks, 6 months
Arm/Group | Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT02640716/Prot_SAP_000.pdf